CLINICAL TRIAL: NCT06823531
Title: Prevalence of Temporomandibular Joint Disorders in Wind Musicians and Their Relationship with Instrument Type
Brief Title: Prevalence of Temporomandibular Joint Disorders in Wind Musicians
Acronym: TMD-WIND
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Maria Blanco Diaz, PhD., University of Oviedo
Other Study IDs: CEIM 795
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: Temporomandibular disorders; TMD; Orofacial pain; Embouchure Disorders; Bruxism; Mandibular Mobility; Jaw diseases
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain; Bruxism; Jaw Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Wind Woodwind Musicians: Musicians playing woodwind instruments (clarinet, saxophone, oboe, fagot, flute).
  Interventions: Other: Not applicable (Observational Study)
- Wind Brass Musicians: Musicians playing brass instruments (trumpet, trombone, tuba, horn).
  Interventions: Other: Not applicable (Observational Study)

INTERVENTIONS:
Other: Not applicable (Observational Study) — Not applicable (Observational Study)

SUMMARY:
This study aims to analyze the prevalence of temporomandibular joint disorders (TMD) in wind musicians, differentiating the impact by instrument type (woodwind vs. brass) and identifying potential risk factors (embouchure, posture, practice time). A cross-sectional observational design will be used, including professional and student musicians from orchestras and conservatories.

DETAILED DESCRIPTION:
This observational cross-sectional study aims to assess the prevalence of temporomandibular joint disorders (TMD) in wind musicians and analyze the impact of instrument type (woodwind vs. brass) on TMD prevalence. Additionally, the study will explore potential risk factors such as embouchure, posture, and practice time.

The study will recruit professional and student wind musicians from orchestras and conservatories. Participants will complete a validated questionnaire (DC/TMD) and undergo a clinical assessment to evaluate mandibular mobility, the presence of joint sounds (clicking, crepitus), and symptoms related to TMD.

The data collection will take place in a single session per participant, estimated between March 1, 2025, and April 15, 2025. The collected data will be analyzed to compare TMD prevalence between different instrument groups and assess correlations with practice habits and postural factors.

All data will be anonymized and stored securely according to applicable data protection regulations (LOPD 3/2018, GDPR 2016/679). Participation in the study is voluntary, and written informed consent will be obtained from all participants, or from their legal guardians in the case of minors.

ELIGIBILITY:
Inclusion Criteria:

* Wind musicians (professional or student).
* Any age (if under 18, parental/legal guardian consent is required).
* Signed informed consent.

Exclusion Criteria:

* History of maxillofacial surgery.
* Presence of neurological disorders affecting mandibular function.
* Recent treatment for TMD.
* Severe bruxism diagnosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of professional and student wind musicians from different orchestras and conservatories. Participants play either woodwind or brass instruments and will be assessed for the prevalence of temporomandibular joint disorders (TMD) and related risk factors. The study includes musicians of any age, with parental consent required for minors.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Temporomandibular Joint Disorders (TMD) in Wind Musicians | Data will be collected in a single session per participant during the study period, estimated from March 1, 2025, to April 15, 2025.
  Percentage of musicians diagnosed with TMD based on the DC/TMD questionnaire and clinical examination.

SECONDARY OUTCOMES:
Comparison of TMD prevalence between woodwind and brass musicians | Data will be collected in a single session per participant during the study period, estimated from March 1, 2025, to April 15, 2025.
  Analysis of differences in TMD prevalence between musicians playing woodwind vs. brass instruments.
Association between practice hours per week and TMD symptoms | Data will be collected in a single session per participant during the study period, estimated from March 1, 2025, to April 15, 2025.
  Exploration of the correlation between weekly practice time and severity of TMD symptoms based on questionnaire responses.
Mandibular Mobility Comparison in Musicians with and without TMD | Data will be collected in a single session per participant during the study period, estimated from March 1, 2025, to April 15, 2025.
  Assessment of differences in maximal mouth opening and mandibular deviation between musicians with and without TMD. Mandibular mobility will be measured using a digital caliper to assess maximal mouth opening (in millimeters) and mandibular deviation. These measurements will be compared between participants diagnosed with TMD and those without TMD